CLINICAL TRIAL: NCT04433572
Title: Temsirolimus Adventitial Delivery to Improve ANGioplasty and/or Atherectomy Revascularization Outcomes Below the Knee: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Effect of Temsirolimus Perivascular Injection 0.1 mg/mL on the Incidence of Ischemia-Driven Major Amputation, Clinically Driven Target Lesion Revascularization, and Clinically Relevant Target Lesion Occlusion After Revascularization of Lesions Below the Knee in Patients With Symptomatic Rutherford 3-5 Peripheral Artery Disease
Brief Title: Temsirolimus Adventitial Delivery to Improve ANGioplasty and/or Atherectomy Revascularization Outcomes Below the Knee
Acronym: TANGO-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mercator MedSystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIP0216
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Artery Disease; Critical Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia | interventions — temsirolimus

STUDY DESIGN:
Intervention Model Description: Block randomization will be stratified for Rutherford 3 and for Rutherford 4/5 participants such that each strata will be randomized 2:1. Block randomization will also be stratified by site such that each site will be assigned a 2:1 randomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The active and placebo material provided to the operator in a blinded syringe or vial will be identical in size, color and appearance. Investigators and participants will be blinded to assignment. Any stents will be placed only after randomization, assignment, and adventitial drug therapy, although any stenting decisions (other than for treatment of AEs) must be made prior to randomization and adventitial drug delivery in order to avoid bias toward or against stenting.
  Participants will not be told of their treatment assignment until after they complete the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Temsirolimus (Active Comparator): Temsirolimus delivered to adventitia and perivascular tissue after primary revascularization
  Interventions: Drug: Temsirolimus
- Placebo (Placebo Comparator): Saline placebo delivered to adventitia and perivascular tissue after primary revascularization
  Interventions: Drug: Saline placebo

INTERVENTIONS:
Drug: Temsirolimus — 0.1 mg/mL temsirolimus, including contrast medium with approximately 75 mg iodine per mL. The dosage will be delivered in a volume of 0.50 mL per cm of target lesion length, up to 30 cm, with +50% allowance for anatomical considerations; for a total volume of up to 22.5 mL and a total dose of up to 2.25 mg in participants assigned to treatment. The same volumes of comparator agent will be delivered in control participants.
  Arms: Temsirolimus
Drug: Saline placebo — Saline placebo, including contrast medium with approximately 75 mg iodine per mL. The dosage will be delivered in a volume of 0.50 mL per cm of target lesion length, up to 30 cm, with +50% allowance for anatomical considerations; for a total volume of up to 22.5 mL and a total dose of up to 2.25 mg in participants assigned to treatment. The same volumes of comparator agent will be delivered in control participants.
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled trial to evaluate the effect of Temsirolimus Perivascular Injection 0.1 mg/mL on the incidence of ischemia-driven major amputation, clinically driven target lesion revascularization, and clinically relevant target lesion occlusion after revascularization of lesions below the knee in patients with symptomatic Rutherford 3-5 peripheral artery disease. The primary safety endpoint will be gathered at 1-month post-index procedure. The primary efficacy endpoint will be gathered at 6 months post-index procedure. Participants will be followed for up to 5 years post-index procedure.

DETAILED DESCRIPTION:
After completion of revascularization therapy and any decision to place stents, participants will be qualified for final enrollment in the study and will be randomized 2:1 and treated with the investigational drug or placebo, respectively. Any stents will be placed only after randomization, assignment, and adventitial drug therapy, although any stenting decisions (other than for treatment of AEs) must be made prior to randomization and adventitial drug delivery in order to avoid bias toward or against stenting.

ELIGIBILITY:
Inclusion Criteria

Pre-procedural:

1. Participant has signed and dated informed consent, is capable of understanding the nature, significance and implications of the clinical trial, and is willing to comply with all study procedures and follow-up visits for the duration of the study.
2. Participant is male or female, aged 18 years or older.
3. If participant is female and of reproductive potential: agreement to use a highly effective contraception (abstinence is acceptable) for at least 90 days after study treatment.
4. Participant has severe claudication (Rutherford 3) or chronic limb-threatening ischemia (CLTI) (Rutherford 4-5) in the Target Limb.

   Angiographic/Procedural:
5. Participant has up to two de novo or restenotic Qualified Target Lesions meeting the following criteria, each based on the Investigator's visual assessment. Target Lesions should be considered separate if they are located in separate vessels (not in the same blood path) or have more than 10 cm intervening normal artery.

   Diameter
   1. ≥70% diameter stenosis anywhere within the Target Lesion or ≥50% diameter stenosis spanning at least 10 cm of length.
   2. Reference (normal) vessel diameter ≥2 mm and ≤8 mm. Location
   3. Any lesion chosen as a Target Lesion is in or spans at least one below-knee popliteal (P3 segment), tibial, or peroneal artery and is a culprit for dominant disease symptoms based on Investigator's assessment.
   4. ≥50% of the Target Lesion length is below the knee joint space (<50% of Target Lesion length may extend above the midline of the knee joint space).
   5. ≥10 mm away from any previously placed stent or graft.
   6. A Target Lesion may cross an ostium of another artery (i.e. pass a bifurcation) but may only include one of the two branches. (Notes: Investigator should choose the dominant lesion for Target Lesion. Bifurcated lesions should be excluded, but if a lesion in a bifurcating vessel is separate from a Target Lesion based on intervening normal artery from which a proximal reference diameter can be measured, it may be treated as a second Target Lesion.) Length
   7. ≤30 cm in cumulative length from most proximal to most distal normal segment bounding the Target Lesion(s).
   8. A single Target Lesion may be comprised of multiple lesions or multifocal lesions (i.e. tandem lesions) if there is no continuous normal segment >10cm in length within the Target Lesion.
   9. Target Lesion may be in a vessel with another Target Lesion or above-knee non-target lesion if it is >10 cm away.
6. Participant receives successful revascularization, based on the following Investigator visual assessments:

   1. Target Lesion and any treated non-target lesion in a Target Vessel or its inflow has <30% residual stenosis, outflow has <50% stenosis, and there is no flow-limiting dissection or perforation after treatment in an inflow vessel or Target Vessel.
   2. Participant has distal run-off into the foot with a patent named pedal artery.

Exclusion Criteria

Pre-procedural:

1. Participant is already enrolled in another clinical study of systemic or local vascular drug therapy or a vascular device study that has not completed its primary endpoint, including prior enrollment in this study.
2. Participant is pregnant, nursing, or planning to become pregnant during the first 12 months after their enrollment in the study.
3. Participant has presence of another anatomic or comorbid condition, or other medical, social, or psychological condition that, in the investigator's opinion, could limit the participant's ability to complete the clinical investigation or comply with follow-up requirements.
4. Incapacitated individuals, defined as persons who are mentally ill, mentally handicapped, or individuals without legal authority, are excluded from the study population.
5. Participant has a life expectancy of ≤1 year.
6. Participant received in the prior 2 months, is currently receiving, or is planned to receive systemic immunosuppressive therapy, immunotherapy or chemotherapy.
7. Participant has platelet count < 100,000 cells per microliter or > 700,000 cells per microliter, or hemoglobin < 7.5 g/dL.
8. Participant is unable to receive H1 antihistamine, temsirolimus or iodinated contrast medium due to labeled contra-indications or known sensitivity reactions except for contrast allergies for which adequate prophylaxis may be used.
9. Participant has a CNS tumor.
10. Participant has had a myocardial infarction within the 30 days prior to study procedure.
11. Participant has had a cerebrovascular accident within the 90 days prior to the study procedure.
12. Participant has had an intracerebral hemorrhage within the 1 year prior to the study procedure.
13. Participant has had any vascular surgical or endovascular procedure performed within the 30 days prior to the Index Procedure or planned within the 30 days after the Index Procedure; allowable exceptions to this exclusion include the following:

    1. Procedures performed during the same setting as the Index Procedure.
    2. Prior staged revascularization in the Target Limb but not the Target Lesion (e.g. for inflow revascularization) within the 30 days prior to the Index Procedure.
14. Participant has a patent, previously implanted bypass graft within 3 cm of the Target Lesion.
15. Participant is bedridden or unable to walk (with assistance is acceptable). Participants in wheelchair who are able to mobilize on their own can be enrolled.
16. Participant has a planned major (above the ankle) amputation in the Target Limb.
17. Participant has had any amputation to the ipsilateral extremity other than the toe or forefoot, or has had major amputation to the contralateral extremity < 1 year prior to index procedure and is not independently ambulating.
18. Participant has signs or symptoms of advanced limb infection or septicemia (fever > 38.5℃, white blood cell count > 15,000 cells per microliter, hypotension) at the time of assessment. Osteomyelitis of the phalanges or metatarsal heads or cellulitis of the foot amenable to treatment with IV antibiotics at the time of revascularization is acceptable.
19. Participant has extensive tissue loss salvageable only with complex foot reconstruction or non-traditional amputations (e.g. Chopart or Lisfranc extending more proximal than a traditional transmetatarsal amputation), including any of the following conditions:

    1. Osteomyelitis that extends proximal to the metatarsal heads. Osteomyelitis limited to the phalanges or metatarsal heads is acceptable for enrollment.
    2. Any of the following involving the plantar skin of the forefoot, midfoot, or heel that cannot be effectively removed with a transmetatarsal amputation:

    i) Gangrene. ii) Deep ulcer (penetrating deeper than the dermis to subcutaneous structures involving facia, muscle or tendon).

    iii) Large shallow ulcer (not penetrating deeper than the dermis and >3cm in any measurement).

    c) Full thickness heel ulcer with or without calcaneal involvement. d) Any wound with calcaneal bone involvement. e) Dorsal wound with extensive necrosis requiring planned amputation more proximal than a transmetatarsal amputation.

    f) Wounds that are deemed to be neuropathic or non-ischemic in nature. g) Wounds that would require flap coverage or complex wound management for large soft tissue defect.
20. Participant has a bilirubin level of >1.5xULN (upper limit of normal range).
21. Participant has an estimated glomerular filtration rate (eGFR) less than 30 mL/min, except for patients with end stage renal disease on stable, chronic dialysis.

    Angiographic/Procedural:
22. Participant has severe, advanced atherosclerotic peripheral artery disease (treated or left untreated) in the Target Limb which, in the opinion of the Investigator, has limited likelihood of a successful outcome.
23. Participant has stenotic lesions, flow limiting dissection, or complication in any of the inflow or outflow vessels in the flow path of the Target Lesion, left untreated or after treatment, with residual stenosis >30% based on the Investigator's visual assessment.
24. Participant receives or has received external radiation therapy to the target limb, vascular brachytherapy, cryotherapy, or drug-coated balloon (DCB) as part of the Target Lesion treatment during the index procedure or previous 6 months.
25. Participant has been treated with a non-resorbable stent/scaffold in the Target Lesion in a prior setting (i.e. in-stent restenosis) or a bioresorbable scaffold in the Target Lesion in the previous 12 months.
26. Participant has a severe (Type C or worse) dissection within the Target Lesion after revascularization but prior to Bullfrog drug delivery.
27. Participant has an untreated aneurysm in the iliac, common femoral, superficial femoral, popliteal, or Target Vessel of the ipsilateral limb.
28. Participant has visible thrombus requiring thrombolysis, percutaneous thrombectomy, or other treatment for acute limb ischemia of the Target Limb.
29. Participant has angiographic evidence of thromboembolism or atheroembolism in the ipsilateral extremity upon completion of the intervention. (Pre- and post-angiographic imaging must confirm the absence of emboli in the distal anatomy.)
30. Participant has a Target Lesion that cannot be crossed with a guide wire; however, subintimal wire crossing is allowed.
31. Participant has heavy calcification at Target Lesion, which in the judgment of the investigator would prevent penetration of the Micro-Infusion Device needle through the vessel wall across the majority of the Target Lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2032-08-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from Cinical Relevant Target Lesion Failure | 6 Months
  Superiority of treatment vs. control group in the composite freedom from the following:
  * Clinically Relevant Target Lesion Occlusion
  * Clinically Driven Target Lesion Revascularization
  * Ischemia-Driven Major Amputation of the Target Limb
MALE + POD | 30 Days
  Noninferiority of treatment vs. control groups in the composite freedom from Major Adverse Limb Event (MALE) in the target limb or Perioperative Death (POD)

SECONDARY OUTCOMES:
Rate of clinically relevant restenosis (CRR) | 6 months
  Superiority of treatment vs. control group in the rate of clinically relevant restenosis (CRR)
Freedom from target lesion failure (TLF) | 6 Months
  Superiority of treatment vs. control group in the composite freedom from the following:
  * Target Lesion Occlusion
  * Clinically Driven Target Lesion Revascularization
  * Ischemia-Driven Major Amputation of the target limb
Freedom from clinically relevant target lesion failure (CR-TLF) | 12 Months
  Superiority of treatment vs. control group in the composite freedom from the following:
  * Clinically Relevant Target Lesion Occlusion
  * Clinically Driven Target Lesion Revascularization
  * Ischemia-Driven Major Amputation of the target limb
Rate of clinically relevant restenosis (CRR) | 12 months
  Superiority of treatment vs. control group in the rate of clinically relevant restenosis (CRR)

OTHER OUTCOMES:
Safety and tolerability will be assessed from overall rate of adverse events (subclassified as major, serious, non-serious, unanticipated, revascularization procedure-related, device-related and drug-related). | 1, 6, 12, 24 months
  AEs/ARs will be categorized into one of the following:
  * MALE of the target limb
  * Non-MALE target limb SAE/SAR
  * Other SAE/SAR
  * Non-serious AE/AR
  AEs/ARs will further be classified as:
  * Expected
  * UADE
  * SUSAR
  AEs/ARs will also be classified for relatedness (definitely, probably, possibly or not) to the following:
  * Revascularization procedure
  * Use of the Bullfrog device
  * The study drug
Freedom from target lesion failure metrics | 1, 6, 12 and 24 months
  Individual endpoints measuring each of the following:
  * Freedom from clinically relevant target lesion failure (CR-TLF)
  * Freedom from target lesion failure (TLF)
  * Freedom from clinically relevant target lesion occlusion (CR-TLO)
  * Freedom from any target lesion occlusion (TLO)
  * Freedom from clinically relevant restenosis (CRR) of the target lesion
Freedom from MALE of the index limb and all-cause death | 1, 6, 12, 24 months
  In composite and separately, the following will be measured:
  * MALE of the index limb
  * All-cause death
Long-term freedom from all-cause death | 36, 48, 60 months
  Rate of freedom from all-cause death
Limb salvage | 1, 6, 12, 24 months
  Freedom from ischemia-driven major amputation
Amputation-free survival | 1, 6, 12, 24 months
  Freedom from ischemia-driven major amputation of the target limb and all-cause death
Thrombotic and embolic outcomes | 1, 6, 12, 24 months
  Examined separately:
  * Arterial thrombosis in the target limb
  * Peripheral embolization in the target limb
  * Acute limb ischemia in the target limb
Patency rates | 1, 6, 12, 24 months
  Examined separately:
  * Primary patency rate
  * Primary assisted patency rate
  * Secondary patency rate
Revascularization rates | 1, 6, 12, 24 months
  Examined separately:
  * Clinically driven target lesion revascularization (CD-TLR)
  * Clinically driven target vessel revascularization (CD-TVR)
  * Clinically driven target vessel revascularization distal to the target lesion
  * Clinically driven target vessel revascularization proximal to the target lesion
Wound healing measures | 1, 6, 12, 24 months
  Examined separately:
  * Index wound assessment for healing
  * Index wound assessment for infection
  * Occurrence of new wound
  * Unassisted wound healing
Rutherford score improvement | 1, 6, 12, 24 months
  Rutherford category and change from baseline
WIfI score improvement | 1, 6, 12, 24 months
  WIfI category and change from baseline
Primary and secondary sustained clinical improvement rates | 1, 6, 12, 24 months
  * Primary sustained clinical improvement rate
  * Secondary sustained clinical improvement rate
Patient reported quality of life benefits (VascuQoL) | 1, 6, 12, 24 months
  VascuQoL results and change from baseline
Patient reported outcomes (walking impairment questionnaire) benefits | 1, 6, 12, 24 months
  WIQ results and change from baseline

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cardiovascular Institute of the South, Houma, Louisiana
  - UT Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
No, there is not a plan to make individual participant data available to other researchers.